CLINICAL TRIAL: NCT00092209
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel Study of the Anti-Hypertensive Efficacy and Safety of Losartan Monotherapy as Compared to HCTZ Monotherapy and to the Combination of Losartan and HCTZ in Japanese Patients With Essential Hypertension
Brief Title: Antihypertensive Efficacy and Safety of Approved Drugs in Japanese Patients With Essential Hypertension (Banyu Study)(0954A-302)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954A-302; 2004_065
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0954A, hydrochlorothiazide (+) losartan potassium
Drug: Comparator: placebo, losartan, hydrochlorothiazide

SUMMARY:
The purpose of this study is to evaluate antihypertensive (lowering blood pressure) effectiveness of three combinations of approved study drugs compared to both study drugs being given alone.

DETAILED DESCRIPTION:
The duration of treatment is 3.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Japanese ancestry
* Stable high blood pressure defined by the study criteria

Exclusion Criteria:

* Pregnant or nursing
* Significant concurrent kidney, liver, blood, or other disease
* Recent heart attack or heart surgery
* History of stroke, severe hypertension (high blood pressure), significant heart failure or cardiac arrhythmias
* Significant lab abnormalities
* Uncontrolled blood sugar
* History of certain drug allergies

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840
Dates: Start 2002-04; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Mean trough SiDBP after 8 weeks of treatment

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Saruta T, Ogihara T, Matsuoka H, Suzuki H, Toki M, Hirayama Y, Nonaka K, Takahashi K. Antihypertensive efficacy and safety of fixed-dose combination therapy with losartan plus hydrochlorothiazide in Japanese patients with essential hypertension. Hypertens Res. 2007 Aug;30(8):729-39. doi: 10.1291/hypres.30.729. PMID 17917321